CLINICAL TRIAL: NCT00281762
Title: Urinary Aquaporin 2 Excretion After NSAID in Fasting Healthy Human
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: MED.RES.HOS.2005.01.TGK
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Healthy
Keywords: AQP-2; NSAID; Urinary concentrating ability
MeSH Terms: interventions — Anti-Inflammatory Agents, Non-Steroidal

INTERVENTIONS:
Drug: NSAID

SUMMARY:
We wanted to test the hypothesis that prostaglandin inhibition reduces the down regulation of u-AQP-2 induced by fasting

ELIGIBILITY:
Inclusion Criteria:

* (1) Genders; both mal and female
* (2) Age; 18- 65 years old
* (3) BMI; below 30
* (4) Females had to bee in oral contraceptive treatment

Exclusion Criteria:

* (1) Clinical signs or history of disease in the heart, lungs, kidneys or endocrine organs
* (2) Abnormal laboratory test (blood haemoglobin, white cell count, platelets, plasma sodium, plasma potassium, plasma creatinine, plasma albumin, plasma bilirubin, plasma alanine aminotransferase, plasma cholesterol and blood glucose)
* (3) Albuminuria or glucosuria
* (4) Cancer
* (5) Arterial hypertension
* (6) Alcohol abuse
* (7) Use of tobacco
* (8) Medical treatment, except oral contraceptives
* (9) Pregnancy or breast feeding
* (10) Medicine abuse
* (11) Donation of blood less than 1 month before the study.

Ages: 18 Years to 65 Years | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
FeNa
U-AQP-2

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Chair — Regional Hospital Holstebro; Thomas G Knudsen, MD, Principal Investigator — Regional Hospital Holstebro
Locations (1):
- Department of Medicine, Holstebro Hospital, Holstebro, Denmark

REFERENCES:
- [Derived] Lauridsen TG, Vase H, Starklint J, Graffe CC, Bech JN, Nielsen S, Pedersen EB. Increased renal sodium absorption by inhibition of prostaglandin synthesis during fasting in healthy man. A possible role of the epithelial sodium channels. BMC Nephrol. 2010 Oct 28;11:28. doi: 10.1186/1471-2369-11-28. PMID 21029429